CLINICAL TRIAL: NCT03245515
Title: Pharmacokinetics and Metabolism of [14C] BMS-986195 in Healthy Male Subjects
Brief Title: A Study of BMS-986195 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM014-016; 2017-002706-12 (EudraCT Number)
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — branebrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BMS-986195 (Experimental): A single oral solution dose of BMS-986195
  Interventions: Drug: BMS-986195

INTERVENTIONS:
Drug: BMS-986195 — specified dose on specified days

SUMMARY:
The purpose of this study is to investigate the effects BMS-986195 in healthy male subjects.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male subjects, if not surgically sterilized, must agree to use adequate contraception
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive (BMI = weight [kg]/[height (m)]2), and total body weight >50 kg
* All prescribed medication, including live vaccinations, must have been stopped at least 30 days prior to admission to the clinical research center
* All over-the-counter (OTC ) medication, vitamin preparations and other food supplements, or herbal medications (eg, St. John's Wort) must have been stopped at least 14 days prior to admission to the clinical research center
* Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks), and grapefruit (juice) from 3 days prior to admission to the clinical research center
* Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, ECG and vital signs, as judged by the Principal Investigator

Exclusion Criteria:

* Previous participation in the current study
* Known previous exposure to BMS-986195
* Employee of PRA or the Sponsor
* History of relevant drug and/or food allergies, including allergy to immunologic or related compounds or allergy to seafood or marine products
* Using tobacco products within 60 days prior to drug administration
* Positive screen for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies or anti-human immunodeficiency virus (HIV) 1 and 2 antibodies

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 16 days
Time to attain maximum observed plasma concentration (tmax) | Up to 16 days
Area under the plasma concentration-time curve up to time t, where t is the last point with concentrations above the lower limit of quantitation [AUC(t-0)] | Up to 16 days
Area under the plasma concentration-time curve from time 0 to infinity calculated as: AUC0-inf = AUC0-t + Ĉlast/kel [AUC(0-inf)] | Up to 16 days
Percentage of estimated part for the calculation of AUC0-inf (%AUCextra) | Up to 16 days
Terminal elimination rate constant (kel) | Up to 16 days
Terminal elimination half life, calculated as 0.693/kel (t1/2) | Up to 16 days
Apparent oral clearance, calculated as dose/AUC0-inf (CL/F) | Up to 16 days
Apparent volume of distribution at terminal phase (Vz/F) | Up to 16 days
Ratio of AUC0-inf of BMS-986195 relative to total radioactivity (TRA) (%) | Up to 16 days
Ratio of AUC0-inf of plasma TRA relative to blood TRA (%) | Up to 16 days
Cumulative amount of TRA excreted in urine (Aeurine) | Up to 16 days
Cumulative amount of TRA excreted in feces (Aefeces) | Up to 16 days
Cumulative amount of TRA excreted in bile (Aebile) | Up to 16 days
Total amount of TRA excreted, calculated as Aetotal = Aeurine + Aefeces | Up to 16 days
Fraction of the dose administered excreted in urine (feurine) | Up to 16 days
Fraction of the dose administered excreted in feces (fefeces) | Up to 16 days
Fraction of the dose administered excreted in bile (febile) | Up to 16 days
Fraction of the dose administered excreted in urine and feces (fetotal) | Up to 16 days

SECONDARY OUTCOMES:
Number of adverse events (AE) | Up to 16 days
Number of serious adverse events (SAE) | Up to 16 days
Number of laboratory test result abnormalities | Up to 16 days
Heart rate measured by ECG | Up to 16 days
PR-interval measured by ECG | Up to 16 days
QRS-duration measured by ECG | Up to 16 days
QT-interval measured by ECG | Up to 16 days
QTc-interval (Fridericia's) measured by ECG | Up to 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Groningen, Netherlands

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx